CLINICAL TRIAL: NCT00327509
Title: Messenger Ribonucleic Acid Expression in Lymphocytes of Glaucoma Patients
Brief Title: mRNA Expression in Lymphocytes of Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Bonn (Other)
Responsible Party: Selim Orgul, University Hospital, Basel, Switzerland
Other Study IDs: 004-KAR-2004-001
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Glaucoma; Healthy Subjects
Keywords: mRNA; glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1-HTG: high tension glaucoma highest IOP > 21 mmHg
- 2-NTG: normal tension glaucoma highest measured IOP < 21 mmHg
- 3-PEX: pseudoexfoliation glaucoma PEX material visible
- 4-Juvenile: juvenile glaucoma
- 5-Control1: healthy subjects (age group 1)
- 6-Control2: healthy subjects (age group 2)

SUMMARY:
The aim of the study is to compare messenger ribonucleic acid (mRNA) expression of various genes in lymphocytes between glaucoma patients and sex and age-matched healthy subjects. A secondary objective is to analyze the impact of different forms of glaucoma or of a vasospastic propensity on the findings.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of blindness world-wide. Chronic primary open-angle glaucoma is the most common form among Caucasian patients. The glaucoma patients will be divided into four groups: (1) high tension glaucoma, (2) normal tension glaucoma, (3) pseudoexfoliation glaucoma, and (4) juvenile glaucoma. Healthy subjects are separated into two age groups. Vasospastic propensity will be assessed with a questionnaire: patients and subjects answering yes to the questions: "do you have always cold hands, even during summer time?" and "do other people tell you that you have cold hands?" will be classified as vasospastic, and as normals if they deny a history of cold hands. Blood will be drawn from an arm vein, lymphocytes will be isolated and mRNA of following genes will be assessed in these lymphocytes:

Nuclear proteins: NF-kappa B, XPGC, P53, XIAP; Multi-drug resistance proteins: ABC 1, ABC 8, MDR 3; Adhesion protein: ICAM 1; Blood brain barrier breakdown protein: P2Y; Energy metabolism proteins: Adrenodoxin, Adrenodoxin-reductase, Cytochrome p450, Cytochrome-reductase, Alcohol-dehydrogenase; Tissue remodeling proteins: MMP 9, MMP 8, MMP 14, TIMP 1, TIMP 2, TIMP 3, TIMP 4.

ELIGIBILITY:
Inclusion Criteria:

Glaucoma patients

* diagnosis of chronic glaucoma with typical glaucomatous disc and visual field damage
* a present or past diurnal tension curve with an average intraocular pressure above 21 mmHg without treatment HTG)
* a present or past diurnal tension curve with an average intraocular pressure below 21 mmHg without treatment (NTG)
* a present or past diurnal tension curve with an average intraocular pressure above 21 mmHg without treatment and signs of pseudoexfoliation in the anterior segment (PEX)
* a juvenile-onset open-angle glaucoma with a present or past diurnal tension curve with an average intraocular pressure above 21 mmHg without treatment (Juvenile Glaucoma)

Healthy subjects

* no history of ocular disease
* no history of systemic disease
* no history of alcohol/drug abuse
* normal blood pressure (100-140 / 60-90 mmHg)
* best corrected visual acuity above 20/25 in both eyes
* no pathological findings upon a slit-lamp examination and indirect fundoscopy
* IOP < 20 mmHg in both eyes

Exclusion Criteria:

* Ametropia > 3 dpt
* Iridocorneal angle extremely narrow with complete or partial closure as determined by gonioscopy
* Pigmentary dispersion
* any abnormality which in the physician's view would prevent reliable applanation tonometry
* History of chronic or recurrent severe inflammatory eye disease such as scleritis or uveitis
* History of ocular trauma or intraocular surgery within the past 6 months
* History of infection or inflammation within the past 3 months
* History of clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy or retinal detachment
* Need for any concomitant medications that may interfere with the evaluation of ocular blood flow
* significant history and/or active alcohol or drug abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: glaucoma patients, healthy subjects
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Eye Clinic, Basel, Canton of Basel-City, Switzerland